CLINICAL TRIAL: NCT02783664
Title: Evaluating the Effects of Genetic Testing on Patients' Stress Levels
Status: Active, not recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Amanda Kong, Associate Professor, Department of Surgery, Division of Surgical Oncology, Medical College of Wisconsin
Other Study IDs: PRO26596
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; BRCA1; BRCA2; stress; gene testing; genetic screening; psychological support; State-Trait Anxiety Inventory; Cancer Worry Scale; Health Anxiety Inventory; gene mutations
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionnaires to Evaluate Patient Stress Levels
  Interventions: Other: Questionnaires to Evaluate Anxiety Related to Genetic Testing

INTERVENTIONS:
Other: Questionnaires to Evaluate Anxiety Related to Genetic Testing — A health team member will outline the study parameters to the patient prior to the genetic counseling visit.
  Visit 1: At the genetic counseling appointment (prior to counseling) patients will receive the following: the State-Trait Anxiety Inventory (STAI) for Adults) to measure baseline anxiety, the Health Anxiety Inventory (HAI) to measure baseline health anxiety, the modified Cancer Worry Scale (CWS) to measure baseline cancer worry in addition to some additional questions about the patient's background. The patient will complete the questionnaires privately and then return them to the genetic counselor.
  Follow-up: One week following disclosure of genetic testing results (3 weeks after the initial appointment), a research team member will call the patient and administer the HAI and CWS over the phone. This will be repeated at 5 weeks, 3 months, and 6 months after initial visit.
  Time to take initial surveys: 15-20 minutes total. Follow-up calls: 10-15 minutes total.

SUMMARY:
This prospective Medical College of Wisconsin Cancer Center study will evaluate stress levels in breast cancer patients undergoing genetic testing. It aims to establish baseline stress levels, evaluate pre- and post-test stress levels at multiple time points, focus on the changes in stress levels for the different resulting subgroups. This will help the clinical staff to provide better care for patients both medically and psychologically through potential interventions to decrease stress.

DETAILED DESCRIPTION:
BACKGROUND: Breast cancer is the second leading cause of cancer death in women (ACS, 2013). Genetic screening has also become increasingly important in treating breast cancer patients, with 5-10% of breast cancers linked to mutations in BRCA1/2 genes(Miki, 1994) (Wooster, 1995). As the field of genetic testing has rapidly expanded and multigene panels are now available, it is unclear what psychological consequences have resulted from the knowledge gained from these tests.

RATIONALE: Breast cancer clinicians frequently employ genetic testing with breast cancer patients. It is unclear what psychological consequences have resulted from the knowledge gained from these tests. A literature review reveals that results are contradictory in terms of determining stress levels related to test results. This is due to different study methodologies. The Medical College of Wisconsin Cancer Center researchers will generate more definitive answers through a prospective study that will establish baseline stress levels, evaluate pre- and post- test stress levels at multiple time points, focus on the changes in stress levels for the different resulting subgroups. Evaluating the impact of genetic testing on stress levels will help health care professionals to better understand the consequences of genetic testing, and thus, provide better care for patients both medically and psychologically through potential interventions to decrease stress.

STUDY PROCEDURES: Patients will be contacted by phone after their genetic counseling appointment is made, prior to their visit by a member of the research team. After giving informed consent, patients will be provided with the State-Trait Anxiety Inventory (STAI) for Adults handout to measure their baseline anxiety, as well as the Health Anxiety Inventory and the Cancer Worry Scale to measure their baseline health anxiety and several additional demographic questions. Subjects will complete the validated questionnaires privately and then return them to the genetic counselor. The data collected at this time point will measure their stress levels before genetic counseling and testing. Patients will be contacted by phone four more times to take the HAI and CWS survey over the phone (one week after receiving genetic testing results, which is three weeks after the consult; at five weeks; three months and six months).

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years or older.
* Identified as currently diagnosed with breast cancer within the past six months or are classified as being at high risk for developing breast cancer (i.e., they have a family history of cancer that puts them at risk for breast cancer) by the Froedtert Hospital & Medical College of Wisconsin Cancer Genetics Screening Program.

Exclusion Criteria:

* Prior genetic testing for breast cancer.
* Patient is a referral for genetic testing from an outside hospital system for whom there is no access to outside medical records.
* Past medical history of breast cancer (not including a current diagnosis of breast cancer within the past six months).
* Current or past history of ovarian cancer.
* Known family history of a BRCA1/2 mutation or cancer susceptibility genetic mutation.
* Patients who are seen in the day hospital for genetic counseling while they are being administered chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Females 18 years or older.
  * Identified as currently diagnosed with breast cancer within the past six months or are classified as being at high risk for developing breast cancer (i.e., they have a family history of cancer that puts them at risk for breast cancer) by the Froedtert Hospital & Medical College of Wisconsin Cancer Genetics Screening Program.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2016-07; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Measure anxiety at baseline using the State-Trait Anxiety Inventory. | Baseline
  The STAI assesses current and trait anxiety symptoms. The investigators use the STAI to measure anxiety at baseline.
Measure change in degree of health anxiety on the questionnaire Health Anxiety Inventory from baseline to six months. | Baseline, 1 Week following results disclosure, 5 Weeks, 3 Months, 6 Months
  Degree of health anxiety measured by the questionnaire Health Anxiety Inventory with 14 and 18-items (HAI). First survey taken at the appointment. Subsequent surveys given over the phone.
Measure change in degree of health anxiety on the questionnaire Cancer Worry Scale from baseline to six months. | Baseline, 1 Week following results disclosure, 5 Weeks, 3 Months, 6 Months
  CWS consists of 6 items and has been used in research to assess concerns about developing cancer or developing cancer again and the impact of these concerns on daily functioning among individuals at risk for hereditary cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Kong, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Cancer Society (ACS). Surveillance and Health Services Research. 2013.
- [Background] Miki Y, Swensen J, Shattuck-Eidens D, Futreal PA, Harshman K, Tavtigian S, Liu Q, Cochran C, Bennett LM, Ding W, et al. A strong candidate for the breast and ovarian cancer susceptibility gene BRCA1. Science. 1994 Oct 7;266(5182):66-71. doi: 10.1126/science.7545954.
- [Background] Wooster R, Bignell G, Lancaster J, Swift S, Seal S, Mangion J, Collins N, Gregory S, Gumbs C, Micklem G. Identification of the breast cancer susceptibility gene BRCA2. Nature. 1995 Dec 21-28;378(6559):789-92. doi: 10.1038/378789a0. PMID 8524414